CLINICAL TRIAL: NCT04084483
Title: A Study Assessing the Safety, Efficacy, and Optimum Dosage of K-161 in Subjects With Moderate to Severe Dry Eye Disease
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Kowa Research Institute, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: K-161-2.01US
Record Dates: First submitted 2019-08-13; First posted 2019-09-10 (Actual); Results first posted 2023-03-15 (Actual); Last update posted 2023-03-15 (Actual); Status verified 2023-02

CONDITIONS: Dry Eye Disease
MeSH Terms: conditions — Dry Eye Syndromes

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (4):
- Group 1 (Experimental): K-161 Ophthalmic Solution Dose A.
  Interventions: Drug: K-161
- Group 2 (Experimental): K-161 Ophthalmic Solution Dose B.
  Interventions: Drug: K-161
- Group 3 (Experimental): K-161 Ophthalmic Solution Dose C.
  Interventions: Drug: K-161
- Group 4 (Placebo Comparator): Vehicle Solution Dose.
  Interventions: Other: Placebo (Vehicle)

INTERVENTIONS:
Drug: K-161 — K-161 alternate dosage
  Arms: Group 1; Group 2; Group 3
Other: Placebo (Vehicle) — Placebo solution
  Arms: Group 4

SUMMARY:
The objective of the study is to assess the safety, efficacy, optimum dosage, and dosing regimen of K-161 in adult subjects with moderate to severe dry eye disease.

ELIGIBILITY:
Inclusion Criteria:

* Be at least 18 years of age at the time of informed consent visit.
* Have a reported history of dry eye disease in both eyes and a history of eye drop use for dry eye symptoms.
* Meet all inclusion criteria outlined in the clinical study protocol.

Exclusion Criteria:

* Have any clinically significant ocular condition.
* Have a history of corneal refractive surgery and/or any other ocular surgical procedure within 12 months.
* Must not meet any other exclusion criteria outlined in the clinical study protocol.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 238 (Actual)
Dates: Start 2019-08-04 (Actual); Primary Completion 2020-01-09 (Actual); Study Completion 2020-01-09 (Actual)

CONTACTS AND LOCATIONS:
Locations (4):
- United States (4):
  - Eye Research Foundation, Newport Beach, California
  - Central Maine Eye Care, Lewiston, Maine
  - Andover Eye Associates, Andover, Massachusetts
  - Total Eye Care, P.A., Memphis, Tennessee

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: During the screening period, two 90-minute exposures to the CAE® were conducted to ascertain eligibility to enter the study. Participants who qualified after the initial screening visit entered the run-in phase, where they self-administered Vehicle for approximately 14 days. Those who qualified at Visit 2 (Day 1) were randomized to receive study drug in a double-masked fashion for 28 days.
Groups:
- Placebo (BID) (Vehicle); 0.025% K-161 (BID); 0.1% K-161 (BID); 0.1% K-161 (QID): 1 drop Ophthalmic Solution
Period: Overall Study
Arm/Group | Placebo (BID) (Vehicle) | 0.025% K-161 (BID) | 0.1% K-161 (BID) | 0.1% K-161 (QID)
Started | 59 | 59 | 61 | 59
Completed | 56 | 57 | 59 | 57
Not Completed | 3 | 2 | 2 | 2

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Placebo (BID) (Vehicle) | 0.025% K-161 (BID) | 0.1% K-161 (BID) | 0.1% K-161 (QID) | Total
Number analyzed (Participants) | 59 | 59 | 61 | 59 | 238
Age, Customized [Count of Participants; unit: Participants]
  < 65 years | 34 | 37 | 38 | 38 | 147
  ≥ 65 years | 25 | 22 | 23 | 21 | 91
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 41 | 43 | 44 | 43 | 171
  Male | 18 | 16 | 17 | 16 | 67
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1 | 1 | 1 | 1 | 4
  Not Hispanic or Latino | 58 | 58 | 60 | 58 | 234
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 1 | 0 | 0 | 0 | 1
  Asian | 13 | 16 | 12 | 15 | 56
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0
  Black or African American | 15 | 11 | 10 | 9 | 45
  White | 29 | 32 | 37 | 35 | 133
  More than one race | 1 | 0 | 2 | 0 | 3
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0
Inferior Corneal Fluorescein Staining Score Post Controlled Adverse Environment (Post-CAE) [Mean (Standard Deviation); unit: scores on a scale] — Fluorescein Staining is measured with the Ora Calibra® Corneal and Conjunctival Staining Scale which is a 0 to 4 scale with increasing half-units and where higher numbers indicating more severe staining. Higher score represents a worsen outcome.
  scores on a scale | 3.30 (0.361) | 3.36 (0.405) | 3.35 (0.412) | 3.33 (0.378) | 3.33 (0.388)
Ocular Discomfort Scale Post-CAE [Mean (Standard Deviation); unit: scores on a scale] — Ocular discomfort scores were subjectively graded by the subjects using the Ora Calibra® Ocular Discomfort Scale from 0 to 4 where 0 = No Discomfort and 4 = Constant Discomfort.
  scores on a scale | 3.8 (0.49) | 3.7 (0.48) | 3.7 (0.61) | 3.6 (0.72) | 3.7 (0.58)

OUTCOME MEASURES:

1. Primary Outcome: Change in Inferior Corneal Fluorescein Staining Score Post Controlled Adverse Environment (Post-Controlled Adverse Environment (CAE))
Description: Fluorescein Staining is measured with the Ora Calibra® Corneal and Conjunctival Staining Scale which is a 0 to 4 scale with increasing half-units and where higher numbers indicating more severe staining.
  K-161 compared to Vehicle. When study patients are exposed to Controlled Adverse Environment (CAE) in terms of relative humidity, temperature, airflow, and visual tasking, the ocular surface is stressed to react. This controlled environmental stress creates a consistent response that's reproducible over time.
Time Frame: Baseline to Day 29
Population: Endpoints analysis was determined by comparing 0.1% K-161 BID to its Vehicle BID
Measure: Least Squares Mean (Standard Error); unit: scores on a scale
Arm/Group | Placebo (BID) (Vehicle) | 0.1% K-161 (BID)
Number analyzed (Participants) | 59 | 61
scores on a scale | -0.57 (0.075) | -0.44 (0.073)
Statistical Analysis 1: Comparison: Placebo (BID) (Vehicle) vs 0.1% K-161 (BID); Test type: Superiority; p = 0.2175, ANCOVA

2. Primary Outcome: Change in Ocular Discomfort Scale Post-CAE
Description: Ocular discomfort scores were subjectively graded by the subjects using the Ora Calibra® Ocular Discomfort Scale from 0 to 4 where 0 = No Discomfort and 4 = Constant Discomfort.
Time Frame: Baseline to Day 29
Population: Endpoints analysis was determined by comparing 0.1% K-161 BID to its Vehicle BID
Measure: Least Squares Mean (Standard Error); unit: score on a scale
Arm/Group | Placebo (BID) (Vehicle) | 0.1% K-161 (BID)
Number analyzed (Participants) | 59 | 61
score on a scale | 0.0 (0.06) | 0.0 (0.06)
Statistical Analysis 1: Comparison: Placebo (BID) (Vehicle) vs 0.1% K-161 (BID); Test type: Superiority; p = 0.3852, ANCOVA

3. Secondary Outcome: Change in Schirmer's Test Value (Unanesthetized) Pre-CAE
Description: Measured with Schirmer's test strip with the length of the moistened area recorded in mm. Lower values indicate less tears produced in the eye.
Time Frame: Baseline to Day 29
Population: Endpoints analysis was determined by comparing 0.1% K-161 BID to its Vehicle BID
Measure: Least Squares Mean (Standard Error); unit: mm
Arm/Group | Placebo (BID) (Vehicle) | 0.1% K-161 (BID)
Number analyzed (Participants) | 59 | 61
mm | 3.4 (0.85) | 2.2 (0.80)
Statistical Analysis 1: Comparison: Placebo (BID) (Vehicle) vs 0.1% K-161 (BID); Test type: Superiority; p = 0.2980, ANCOVA

4. Secondary Outcome: Change in Tear Film Break-up Time (TFBUT) Post-CAE
Time Frame: Baseline to Day 29
Population: Endpoints analysis was determined by comparing 0.1% K-161 BID to its Vehicle BID
Measure: Least Squares Mean (Standard Error); unit: Seconds
Arm/Group | Placebo (BID) (Vehicle) | 0.1% K-161 (BID)
Number analyzed (Participants) | 59 | 61
Seconds | 0.402 (0.1090) | 0.132 (0.1049)
Statistical Analysis 1: Comparison: Placebo (BID) (Vehicle) vs 0.1% K-161 (BID); Test type: Superiority; p = 0.0634, ANCOVA

5. Secondary Outcome: Change in Fluorescein Staining Scores (Pre-CAE®)
Description: Fluorescein Staining is measured with the Ora Calibra® Corneal and Conjunctival Staining Scale which is a 0 to 4 scale with increasing half-units and where higher numbers indicating more severe staining.
Time Frame: Baseline to Day 29
Population: Endpoints analysis was determined by comparing Vehicle BID to 0.1% K-161 BID and 0.025% K-161 BID
Measure: Least Squares Mean (Standard Error); unit: score on a scale
Arm/Group | Placebo (BID) (Vehicle) | 0.025% K-161 (BID) | 0.1% K-161 (BID)
Number analyzed (Participants) | 59 | 59 | 61
score on a scale
  Corneal Sum | -0.28 (0.184) | -0.36 (0.182) | -0.50 (0.178)
  Conjunctival Sum | -0.03 (0.138) | -0.22 (0.136) | -0.28 (0.133)
  Total Eye Sum | -0.30 (0.292) | -0.59 (0.290) | -0.80 (0.283)
Statistical Analysis 1: Comparison: Placebo (BID) (Vehicle) vs 0.025% K-161 (BID); Corneal Sum; Test type: Superiority; p = 0.7388, ANCOVA
Statistical Analysis 2: Comparison: Placebo (BID) (Vehicle) vs 0.1% K-161 (BID); Corneal Sum; Test type: Superiority; p = 0.3717, ANCOVA
Statistical Analysis 3: Comparison: Placebo (BID) (Vehicle) vs 0.025% K-161 (BID); Conjunctival Sum; Test type: Superiority; p = 0.3164, ANCOVA
Statistical Analysis 4: Comparison: Placebo (BID) (Vehicle) vs 0.1% K-161 (BID); Conjunctival Sum; Test type: Superiority; p = 0.1953, ANCOVA
Statistical Analysis 5: Comparison: Placebo (BID) (Vehicle) vs 0.025% K-161 (BID); Total Eye Sum; Test type: Superiority; p = 0.4645, ANCOVA
Statistical Analysis 6: Comparison: Placebo (BID) (Vehicle) vs 0.1% K-161 (BID); Total Eye Sum; Test type: Superiority; p = 0.2135, ANCOVA

6. Secondary Outcome: Change in Lissamine Green Staining (Pre-CAE) Using the Ora Calibra® Scale (Conjunctival Sum)
Description: Ora Calibra Scale which is 0 to 4 scale with increasing half-units and where higher numbers indicating more severe staining.
Time Frame: Baseline to Day 29
Population: Endpoints analysis was determined by comparing Vehicle BID to 0.1% K-161 BID and 0.025% K-161 BID
Measure: Least Squares Mean (Standard Error); unit: score on a scale
Arm/Group | Placebo (BID) (Vehicle) | 0.025% K-161 (BID) | 0.1% K-161 (BID)
Number analyzed (Participants) | 59 | 59 | 61
score on a scale | -0.16 (0.132) | -0.25 (0.131) | -0.39 (0.127)
Statistical Analysis 1: Comparison: Placebo (BID) (Vehicle) vs 0.025% K-161 (BID); Test type: Superiority; p = 0.5990, ANCOVA
Statistical Analysis 2: Comparison: Placebo (BID) (Vehicle) vs 0.1% K-161 (BID); Test type: Superiority; p = 0.2122, ANCOVA

7. Secondary Outcome: Change in Conjunctival Redness (Pre-CAE)
Description: Conjunctival Redness Scale ranges from 0 to 4, where 0 = normal, without vasodilation and 4 = Broad Ciliary and Prominent, Horizontal Conjunctival Vasodilation. Higher scores indicate worsening conjunctival redness.
Time Frame: Baseline to Day 29
Population: Endpoints analysis was determined by comparing Vehicle BID to 0.1% K-161 BID and 0.025% K-161 BID
Measure: Least Squares Mean (Standard Error); unit: Point
Arm/Group | Placebo (BID) (Vehicle) | 0.025% K-161 (BID) | 0.1% K-161 (BID)
Number analyzed (Participants) | 59 | 59 | 61
Point | -0.21 (0.061) | -0.20 (0.060) | -0.22 (0.059)
Statistical Analysis 1: Comparison: Placebo (BID) (Vehicle) vs 0.025% K-161 (BID); Test type: Superiority; p = 0.9146, ANCOVA
Statistical Analysis 2: Comparison: Placebo (BID) (Vehicle) vs 0.1% K-161 (BID); Test type: Superiority; p = 0.8494, ANCOVA

8. Secondary Outcome: Change in Tear Film Break-Up Time (Pre CAE)
Time Frame: Baseline to Day 29
Population: Endpoints analysis was determined by comparing Vehicle BID to 0.1% K-161 BID and 0.025% K-161 BID
Measure: Least Squares Mean (Standard Error); unit: Seconds
Arm/Group | Placebo (BID) (Vehicle) | 0.025% K-161 (BID) | 0.1% K-161 (BID)
Number analyzed (Participants) | 59 | 59 | 61
Seconds | 0.312 (0.0880) | 0.398 (0.0863) | 0.242 (0.0848)
Statistical Analysis 1: Comparison: Placebo (BID) (Vehicle) vs 0.025% K-161 (BID); Test type: Superiority; p = 0.4747, ANCOVA
Statistical Analysis 2: Comparison: Placebo (BID) (Vehicle) vs 0.1% K-161 (BID); Test type: Superiority; p = 0.5619, ANCOVA

9. Secondary Outcome: Change in Tear Osmolarity (Pre CAE)
Time Frame: Baseline to Day 29
Population: Endpoints analysis was determined by comparing Vehicle BID to 0.1% K-161 BID and 0.025% K-161 BID
Measure: Least Squares Mean (Standard Error); unit: mOsm/L
Arm/Group | Placebo (BID) (Vehicle) | 0.025% K-161 (BID) | 0.1% K-161 (BID)
Number analyzed (Participants) | 59 | 59 | 61
mOsm/L | -0.5 (2.17) | 1.0 (2.09) | 0.4 (2.03)
Statistical Analysis 1: Comparison: Placebo (BID) (Vehicle) vs 0.025% K-161 (BID); Test type: Superiority; p = 0.5985, ANCOVA
Statistical Analysis 2: Comparison: Placebo (BID) (Vehicle) vs 0.1% K-161 (BID); Test type: Superiority; p = 0.7626, ANCOVA

10. Secondary Outcome: Change in Unanesthetized Schirmer's Test (Pre CAE)
Description: as for outcome 3
Time Frame: Baseline to Day 29
Population: Endpoints analysis was determined by comparing Vehicle BID to 0.1% K-161 BID and 0.025% K-161 BID
Measure: Least Squares Mean (Standard Error); unit: mm
Arm/Group | Placebo (BID) (Vehicle) | 0.025% K-161 (BID) | 0.1% K-161 (BID)
Number analyzed (Participants) | 59 | 59 | 61
mm | 3.3 (0.82) | 3.1 (0.80) | 2.1 (0.78)
Statistical Analysis 1: Comparison: Placebo (BID) (Vehicle) vs 0.025% K-161 (BID); Test type: Superiority; p = 0.8330, ANCOVA
Statistical Analysis 2: Comparison: Placebo (BID) (Vehicle) vs 0.1% K-161 (BID); Test type: Superiority; p = 0.2777, ANCOVA

11. Secondary Outcome: Change in Blink Rate (Pre CAE)
Description: Blinks per 60 seconds.
Time Frame: Baseline to Day 29
Population: Endpoints analysis was determined by comparing Vehicle BID to 0.1% K-161 BID and 0.025% K-161 BID
Measure: Least Squares Mean (Standard Error); unit: Blinks per 60 seconds
Arm/Group | Placebo (BID) (Vehicle) | 0.025% K-161 (BID) | 0.1% K-161 (BID)
Number analyzed (Participants) | 59 | 59 | 61
Blinks per 60 seconds | 0.1 (1.41) | 0.1 (1.39) | -0.2 (1.36)
Statistical Analysis 1: Comparison: Placebo (BID) (Vehicle) vs 0.025% K-161 (BID); Test type: Superiority; p = 0.9829, ANCOVA
Statistical Analysis 2: Comparison: Placebo (BID) (Vehicle) vs 0.1% K-161 (BID); Test type: Superiority; p = 0.8675, ANCOVA

12. Secondary Outcome: Change in Ocular Discomfort Scale (Pre CAE)
Description: Ora Calibra® Ocular Discomfort Scale ranging from 0 to 4
Time Frame: Baseline to Day 29
Population: Endpoints analysis was determined by comparing Vehicle BID to 0.1% K-161 BID and 0.025% K-161 BID
Measure: Least Squares Mean (Standard Error); unit: Score
Arm/Group | Placebo (BID) (Vehicle) | 0.025% K-161 (BID) | 0.1% K-161 (BID)
Number analyzed (Participants) | 59 | 59 | 61
Score | -0.3 (0.13) | -0.2 (0.13) | -0.5 (0.12)
Statistical Analysis 1: Comparison: Placebo (BID) (Vehicle) vs 0.025% K-161 (BID); Test type: Superiority; p = 0.5836, ANCOVA
Statistical Analysis 2: Comparison: Placebo (BID) (Vehicle) vs 0.1% K-161 (BID); Test type: Superiority; p = 0.2352, ANCOVA

13. Secondary Outcome: Change in Ocular Discomfort and 4-Symptom Questionnaire (Pre CAE)
Description: Scores ranging from 0 to 5. A score of 0 indicates no discomfort/symptoms and a score of 5 indicates worst discomfort/symptoms.
Time Frame: Baseline to Day 29
Population: Endpoints analysis was determined by comparing Vehicle BID to 0.1% K-161 BID and 0.025% K-161 BID
Measure: Least Squares Mean (Standard Error); unit: Point
Arm/Group | Placebo (BID) (Vehicle) | 0.025% K-161 (BID) | 0.1% K-161 (BID)
Number analyzed (Participants) | 59 | 59 | 61
Point
  Ocular Discomfort | -0.2 (0.13) | -0.2 (0.13) | -0.4 (0.13)
  Burning | 0.1 (0.13) | 0.0 (0.13) | -0.1 (0.13)
  Dryness | -0.1 (0.14) | -0.2 (0.14) | -0.3 (0.13)
  Grittiness | -0.1 (0.15) | -0.3 (0.15) | -0.1 (0.15)
  Stinging | -0.1 (0.15) | -0.1 (0.15) | -0.2 (0.14)
Statistical Analysis 1: Comparison: Placebo (BID) (Vehicle) vs 0.025% K-161 (BID); Ocular Discomfort; Test type: Superiority; p = 0.7367, ANCOVA
Statistical Analysis 2: Comparison: Placebo (BID) (Vehicle) vs 0.1% K-161 (BID); Ocular Discomfort; Test type: Superiority; p = 0.3865, ANCOVA
Statistical Analysis 3: Comparison: Placebo (BID) (Vehicle) vs 0.025% K-161 (BID); Burning; Test type: Superiority; p = 0.8796, ANCOVA
Statistical Analysis 4: Comparison: Placebo (BID) (Vehicle) vs 0.1% K-161 (BID); Burning; Test type: Superiority; p = 0.3515, ANCOVA
Statistical Analysis 5: Comparison: Placebo (BID) (Vehicle) vs 0.025% K-161 (BID); Dryness; Test type: Superiority; p = 0.6338, ANCOVA
Statistical Analysis 6: Comparison: Placebo (BID) (Vehicle) vs 0.1% K-161 (BID); Dryness; Test type: Superiority; p = 0.4685, ANCOVA
Statistical Analysis 7: Comparison: Placebo (BID) (Vehicle) vs 0.025% K-161 (BID); Grittiness; Test type: Superiority; p = 0.4757, ANCOVA
Statistical Analysis 8: Comparison: Placebo (BID) (Vehicle) vs 0.1% K-161 (BID); Grittiness; Test type: Superiority; p = 0.8803, ANCOVA
Statistical Analysis 9: Comparison: Placebo (BID) (Vehicle) vs 0.025% K-161 (BID); Stinging; Test type: Superiority; p = 0.8529, ANCOVA
Statistical Analysis 10: Comparison: Placebo (BID) (Vehicle) vs 0.1% K-161 (BID); Stinging; Test type: Superiority; p = 0.7713, ANCOVA

14. Secondary Outcome: Change in Visual Analog Scale (Pre CAE)
Description: The length of the assessment line was 100 mm; a measure of 0 mm corresponded to "no discomfort" and 100 mm corresponds to "maximal discomfort".
Time Frame: Baseline to Day 29
Population: Endpoints analysis was determined by comparing Vehicle BID to 0.1% K-161 BID and 0.025% K-161 BID
Measure: Least Squares Mean (Standard Error); unit: mm
Arm/Group | Placebo (BID) (Vehicle) | 0.025% K-161 (BID) | 0.1% K-161 (BID)
Number analyzed (Participants) | 59 | 59 | 61
mm
  Burning/Stinging | -1.9 (2.78) | -7.6 (2.76) | -5.6 (2.68)
  Itching | -3.1 (2.92) | -9.7 (2.92) | -6.1 (2.84)
  Foreign Body Sensation | -1.1 (2.96) | -6.9 (2.94) | -5.6 (2.82)
  Blurry Vision | -0.2 (2.69) | -5.5 (2.67) | -7.5 (2.60)
  Eye Dryness | -4.1 (2.71) | -6.1 (2.68) | -10.7 (2.60)
  Photophobia | -2.8 (2.78) | -6.2 (2.75) | -10.7 (2.67)
  Pain | 0.0 (2.37) | -6.0 (2.37) | -4.2 (2.28)
Statistical Analysis 1: Comparison: Placebo (BID) (Vehicle) vs 0.025% K-161 (BID); Burning/Stinging; Test type: Superiority; p = 0.1380, ANCOVA
Statistical Analysis 2: Comparison: Placebo (BID) (Vehicle) vs 0.1% K-161 (BID); Burning/Stinging; Test type: Superiority; p = 0.3334, ANCOVA
Statistical Analysis 3: Comparison: Placebo (BID) (Vehicle) vs 0.025% K-161 (BID); Itching; Test type: Superiority; p = 0.1008, ANCOVA
Statistical Analysis 4: Comparison: Placebo (BID) (Vehicle) vs 0.1% K-161 (BID); Itching; Test type: Superiority; p = 0.4582, ANCOVA
Statistical Analysis 5: Comparison: Placebo (BID) (Vehicle) vs 0.025% K-161 (BID); Foreign Body Sensation; Test type: Superiority; p = 0.1511, ANCOVA
Statistical Analysis 6: Comparison: Placebo (BID) (Vehicle) vs 0.1% K-161 (BID); Foreign Body Sensation; Test type: Superiority; p = 0.2555, ANCOVA
Statistical Analysis 7: Comparison: Placebo (BID) (Vehicle) vs 0.025% K-161 (BID); Blurry Vision; Test type: Superiority; p = 0.1546, ANCOVA
Statistical Analysis 8: Comparison: Placebo (BID) (Vehicle) vs 0.1% K-161 (BID); Blurry Vision; Test type: Superiority; p = 0.0495, ANCOVA
Statistical Analysis 9: Comparison: Placebo (BID) (Vehicle) vs 0.025% K-161 (BID); Eye Dryness; Test type: Superiority; p = 0.5791, ANCOVA
Statistical Analysis 10: Comparison: Placebo (BID) (Vehicle) vs 0.1% K-161 (BID); Eye Dryness; Test type: Superiority; p = 0.0736, ANCOVA
Statistical Analysis 11: Comparison: Placebo (BID) (Vehicle) vs 0.025% K-161 (BID); Photophobia; Test type: Superiority; p = 0.3666, ANCOVA
Statistical Analysis 12: Comparison: Placebo (BID) (Vehicle) vs 0.1% K-161 (BID); Photophobia; Test type: Superiority; p = 0.0390, ANCOVA
Statistical Analysis 13: Comparison: Placebo (BID) (Vehicle) vs 0.025% K-161 (BID); Pain; Test type: Superiority; p = 0.0655, ANCOVA
Statistical Analysis 14: Comparison: Placebo (BID) (Vehicle) vs 0.1% K-161 (BID); Pain; Test type: Superiority; p = 0.1947, ANCOVA

15. Secondary Outcome: Change in Ocular Surface Disease Index Score (Pre-CAE) - Total OSDI
Description: The OSDI© is comprised of 12 questions, with each question assessed on a scale ranging from 0 to 4 where 0 = none of the time, 1 = some of the time, 2 = half of the time, 3 = most of the time, and 4 = all of the time. The range of total score is "0 to 100". "Subscale" scores are not reported. Higher score represents a worsen outcome. The total score is the sum of subscales.
Time Frame: Baseline to Day 29
Population: Endpoints analysis was determined by comparing Vehicle BID to 0.1% K-161 BID and 0.025% K-161 BID
Measure: Least Squares Mean (Standard Error); unit: scores on a scale
Arm/Group | Placebo (BID) (Vehicle) | 0.025% K-161 (BID) | 0.1% K-161 (BID)
Number analyzed (Participants) | 59 | 59 | 61
scores on a scale | -3.2 (2.03) | -2.9 (2.00) | -7.8 (1.95)
Statistical Analysis 1: Comparison: Placebo (BID) (Vehicle) vs 0.025% K-161 (BID); Test type: Superiority; p = 0.9274, ANCOVA
Statistical Analysis 2: Comparison: Placebo (BID) (Vehicle) vs 0.1% K-161 (BID); Test type: Superiority; p = 0.0888, ANCOVA

ADVERSE EVENTS:
Time Frame: 36 Days
Description: Treatment emergent adverse events (TEAE) were any adverse event that occurred or worsened after the first dose of study treatment.
Arm/Group | Placebo (BID) (Vehicle) | 0.025% K-161 (BID) | 0.1% K-161 (BID) | 0.1% K-161 (QID)
All-Cause Mortality (participants affected / at risk) | 0/59 | 0/59 | 0/61 | 0/59
Serious Adverse Events (participants affected / at risk) | 3/59 | 0/59 | 0/61 | 0/59
Other Adverse Events (participants affected / at risk) | 2/59 | 7/59 | 25/61 | 24/59
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo (BID) (Vehicle) (N=59) | 0.025% K-161 (BID) (N=59) | 0.1% K-161 (BID) (N=61) | 0.1% K-161 (QID) (N=59)
Pelvic fracture (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0
Upper limb fracture (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0
Pneumonia (Infections and infestations) | 1 | 0 | 0 | 0
Acute kidney injury (Renal and urinary disorders) | 1 | 0 | 0 | 0
Toxic encephalopathy (Nervous system disorders) | 1 | 0 | 0 | 0
Chronic lymphocytic leukaemia (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo (BID) (Vehicle) (N=59) | 0.025% K-161 (BID) (N=59) | 0.1% K-161 (BID) (N=61) | 0.1% K-161 (QID) (N=59)
Instillation site pain (General disorders) | 2 | 6 | 23 | 21 — General disorders and administration site conditions
Dysgeusia (Nervous system disorders) | 0 | 1 | 2 | 3

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes

DOCUMENTS (4):
  • Study Protocol: Protocol (2018-09-14): https://cdn.clinicaltrials.gov/large-docs/83/NCT04084483/Prot_000.pdf
  • Study Protocol: Amendment 1 (2019-06-13): https://cdn.clinicaltrials.gov/large-docs/83/NCT04084483/Prot_001.pdf
  • Study Protocol: Amendment 2 (2019-07-26): https://cdn.clinicaltrials.gov/large-docs/83/NCT04084483/Prot_002.pdf
  • Statistical Analysis Plan (2020-01-03): https://cdn.clinicaltrials.gov/large-docs/83/NCT04084483/SAP_003.pdf